CLINICAL TRIAL: NCT02386631
Title: Hallux Valgus and the Effects of Custom Orthotic Prescription on the Efficacy of Forward Propulsion
Brief Title: Hallux Valgus and Custom Orthotic Prescription
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Stephen Perry (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Perry, Professor, Wilfrid Laurier University
Organization: Wilfrid Laurier University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC_HVFP
Record Dates: First submitted 2015-03-02; First posted 2015-03-12 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Hallux Valgus
Keywords: gait; orthotics; kinetics; hallux valgus; bunions
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orthotic (Experimental): Custom made orthotic provided for study
  Interventions: Device: Custom Made Orthotic

INTERVENTIONS:
Device: Custom Made Orthotic — Provides longitudinal arch support

SUMMARY:
Hallux valgus can be defined as a progressive subluxation of the first metatarsophalangeal joint and lateral deviation of the hallux. This common foot condition is associated with altered gait patterns. Specifically reduced forward propulsion, leading to gait instability. Research has shown that foot problems and pain play a major role towards the contribution of falls in the adult population. There are currently two main interventions for the treatment of hallux valgus: surgery and orthotic prescription. There has not been a lot of research performed evaluating the effects of custom orthotic prescription on hallux valgus.

Therefore, this study will investigate adults with moderate hallux valgus and the effects of orthotic intervention on the efficacy of forward propulsion during walking. It is hypothesized that implementation of an orthotic will lead to decreased foot pain, an increase in step length, an increase in the forward moment about the ankle and hallux, and a more medial center of pressure tracking through the great toe instead of the lesser metatarsals.

This study will consist of 10 adults. The participant will go through three rounds of testing in the lab. The first session will consist of initial baseline testing in which each participant will be evaluated for severity of Hallux Valgus and range of motion of the first metatarsophalangeal joint. A foot casting will then be performed by a pedorthist and the participant will be set up with markers, so as to record motion while they perform 15 walking trials across a 10m runway with a force plate embedded in the middle whilst wearing standard footwear (no orthotic). The second lab session will consist of the standard footwear (no orthotic) walking as well as the addition of standard footwear with custom orthotic walking. The third session, after having worn the orthotic for two weeks, will repeat both conditions measured in the second lab session. Data about the center of pressure trajectories, step length, foot pain, and the moments about the ankle and first metatarsophalangeal joints will be collected and calculated.

DETAILED DESCRIPTION:
The participants will enter the lab three times. On their first session, the level of severity of hallux valgus of the participant will be identified. The participant will sit in a chair, with their bare feet resting on the ground. A picture of their foot will be taken in the transverse plane. Another picture will then be taken of the foot when the individual is in a standing position. The participant will not experience any pain or discomfort during this test as only 2 pictures will be taken of the foot.

The participant will then have range of motion testing performed on their first metatarsophalangeal joint. This will be performed by the researcher passively dorsiflexing the first metatarsophalangeal joint and measuring the angle created with a goniometer.

The participant will also have an orthotic foot casting performed by a pedorthist. This foot casting will be performed to create a mould of the foot that will be used by a pedorthist to construct the orthotic.

After the participant put on the standard footwear (no orthotic) they will be set up with optotrak markers with three on the first ray, three on the midfoot, three on the heel, and three on the medial distal tibia. Then the participant will walk across a 10m walkway with a force plate embedded half way along the walkway at a constant velocity for a total of 15 trials. The participant will rate their pain on the visual analogue scale (VAS) immediately following the completion of the 15 walking trials.

On the second session, the participant will once again be set up with optotrak marker and will perform 15 walking trials with the standard footwear (no orthotics) and rate their pain level on the VAS. The custom orthotic will be placed in the standard footwear. Then the participant will perform 15 walking trials and rate their pain on the VAS. The participant will then be instructed to wear the orthotic for seven hours a day, seven days a week for two weeks. During this two week period, the principal investigator will call the participant once, after about 1 week, to ask about how the orthotic wear is going. In specific, how often they have been wearing it and for how long.

Two weeks later, the participant will return for their final testing session. This session will consist of a repetition of the 15 walking trials and vas ratings with both the standard footwear (no orthotic) and the standard footwear with the custom orthotic. The participant will then be debriefed and offered the opportunity to opt to have a summary of the results when the study is completed sent to them. They will be allowed to keep the custom orthotic.

ELIGIBILITY:
Inclusion Criteria:

* moderate Hallux Valgus, as classified using the Manchester Scale
* good range of motion of the first metatarsophalangeal joint
* able to walk

Exclusion Criteria:

* no history or clinical evidence of any chronic disease and no history of lower extremity surgery
* medication that affect balance and stability

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Increased Propulsive moments (torques) as measured by inverse dynamics | measured at each visit (baseline, 1 week, 2 weeks), orthotic vs. no orthotic
  calculation of moments (torques) produced at the ankle and first metatarsophalangeal joint during push-off phase of the gait cycle

SECONDARY OUTCOMES:
Increased Gait Velocity | measured at each visit (baseline, 1 week, 2 weeks), orthotic vs. no orthotic
  tracking of the individual's center of mass during walking

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Perry, PhD, Study Director — Wilfrid Laurier University
Locations (1):
- WLU Biomechanics Laboratory, Waterloo, Ontario, Canada